CLINICAL TRIAL: NCT05984472
Title: 3-year Clinical Performance of Prefabricated and Clear Template-formed Resin Composite Veneers
Brief Title: 3-year Clinical Performance of Prefabricated and Composite Veneers
Acronym: Edelweiss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sebnem Turkun, Prof. Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-11.1T/15
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Dental Diseases; Tooth Discoloration
Keywords: veneers; anterior restorations; resin composite; prefabricated veneers
MeSH Terms: conditions — Stomatognathic Diseases; Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: Individual Randomized Assignment
Who Masked: Participant, Care Provider
Masking Description: Double (Participant, Evaluator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edelweiss Prefabricated Veneers (Active Comparator): Edelweiss veneers (device 1) were randomly applied to patients. The teeth were evaluated in terms of color and size matching in order to select the correct veneers. Edelweiss sizing guide was used for size selection. Prefabricated veneers were adapted to the teeth' surfaces. Then, the inner surfaces of the prefabricated veneers were roughened to obtain better mechanical retention. Then the labial surfaces of the teeth were etched using 36% phosphoric acid. The etched surfaces were rinsed and dried. An adhesive system was applied to the teeth. Prefabricated veneers' inner surfaces were cleaned with alcohol, and Veneer Bond dental adhesive was applied. Edelweiss nanohybrid resin composite was placed on the inner surfaces of the veneers and transferred to the teeth. These restorations were light-cured for 40 s Gingival borders were adapted with contouring and polishing discs (intervention 1).
  Interventions: Procedure: Edelweiss prefabricated veneers
- Ceram-X Duo SphereTec with U-Veneer (Active Comparator): Direct resin composite restorations were randomly applied to patients. Ceram-X Duo SphereTec resin composite (device 2) was used for color selection. Then U-Veneer transparent templates were tried to select their correct size. After the preparation, the labial surfaces of the teeth were etched using 36% phosphoric acid. The etched surfaces were then rinsed and dried. An adhesive system was applied to the teeth. Then Ceram-X Duo SphereTec nanohybrid resin composite with dentin shade was placed on labial surfaces of teeth and was light-cured. After that Ceram-X Duo SphereTec nanohybrid resin composite enamel shade was placed on the inner surface of the transparent template and was transferred to the tooth. After that, the resin composite veneer was light-cured for 20 s from each surface. The transparent template was removed. Gingival borders were adapted with contouring and polishing discs. Then proximal surfaces were polished using proximal sandpaper strips (intervention 2).
  Interventions: Procedure: Ceram-X Duo SphereTec with U-Veneer

INTERVENTIONS:
Procedure: Edelweiss prefabricated veneers — Individual Randomized Clinical Trial
  Arms: Edelweiss Prefabricated Veneers
Procedure: Ceram-X Duo SphereTec with U-Veneer — Ceram-X Duo SphereTec with U-Veneer
  Arms: Ceram-X Duo SphereTec with U-Veneer

SUMMARY:
The aim of this study was to evaluate the clinical performances of Edelweiss prefabricated veneers and direct resin composite restorations (Ceram-X Duo SphereTec) performed with U- veneer transparent templates used for anterior diastema closure and tooth reshaping over 3-year.

The patient group consisted of individuals who applied for aesthetic complaints on their anterior teeth. 21 volunteer individuals without systemic disease were included in the study. Patients were randomly selected for each group. In Group 1; 38 teeth (10 patients) were restored with Edelweiss prefabricated veneers (Edelweiss Dentistry) in combination with Edelweiss nanohybrid resin composite (Edelweiss Dentistry) and Prime&Bond Universal (Dentsply Sirona) adhesive system. In Group 2; 36 teeth (11 patients) were restored with Ceram-X Duo SphereTec (Dentsply Sirona) resin composite in combination with U- veneer (Ultradent) transparent templates and Prime&Bond Universal adhesive systems. Properties of the restorations were evaluated at baseline, 6, 12, 24, and 36 months using Modified Ryge Criteria (USPHS Criteria). Data were evaluated using Chi-Square and Fisher's Exact tests (p=0.05).

DETAILED DESCRIPTION:
The aim of this study was to evaluate the clinical performances of Edelweiss prefabricated veneers and direct resin composite restorations (Ceram-X Duo SphereTec) performed with U- veneer transparent templates used for anterior diastema closure and tooth reshaping over 3-year.

The study protocol was approved by the Ethical Committee of Ege University, Izmir, Turkey (18-11.1T/15; 28.11.2018). 21 patients (1 male, 20 females, mean age: 35) with aesthetic complaints on their anterior teeth were treated with 74 restorations. 21 volunteer individuals without systemic disease were included in the study. Patients were randomly selected for each group. In Group 1; 38 teeth (10 patients) were restored with Edelweiss prefabricated veneers (Edelweiss Dentistry) in combination with Edelweiss nanohybrid resin composite (Edelweiss Dentistry) and Prime&Bond Universal (Dentsply Sirona) adhesive system. In Group 2; 36 teeth (11 patients) were restored with Ceram-X Duo SphereTec (Dentsply Sirona) resin composite in combination with U- veneer (Ultradent) transparent templates and Prime&Bond Universal adhesive systems.

Periodontal treatments, fillings, and bleaching treatments were performed, if necessary, before any veneer treatment. For the pre-treatment records; 3 photographs (smile, anterior occlusion, and upper anterior teeth alone) were taken from each patient. The "Button Try" technique was used for color selection in both groups. Edelweiss sizing guide was used for size selection in Group 1. U-Veneer (Ultradent) transparent templates were tried on the labial surfaces of teeth to select the correct size in Group 2. Then teeth were cleaned with non-fluoride pumice (Cleanic; Kerr Dental, ABD) using a polishing brush. Isolation of the teeth and retraction of the lips were achieved with a disposable mouth retractor (OptraGate, Ivoclar Vivadent). Prefabricated veneers were prepared for the cementation process in Group 1. Then the labial surfaces were etched using 36% phosphoric acid for 30 s. The etched surfaces were rinsed for 30 s and dried. Prime&Bond Universal (Dentsply Sirona) adhesive system was applied on the labial surfaces of the teeth in accordance with user instructions in both groups. In Group 1; Edelweiss nano hybrid resin composite was placed on the inner surfaces of the prefabricated veneers before being applied on appropriate teeth. Then the restorations were light-cured for 40 s from each surface (D-Light Pro, GC). In Group 2; Ceram-X Duo SphereTec (Dentsply Sirona) nanohybrid resin composite with dentin color was placed on the labial surfaces of the teeth and light-cured (D-Light Pro, GC). After that layer, Ceram-X Duo SphereTec (Dentsply Sirona) enamel shades were placed on the inner surface of the transparent template and pressed against the labial surface of the tooth. After the removal of the excess materials, the resin composite veneer was light-cured for 20 s from each surface. Then the transparent template was removed.

In both groups; gingival borders were adapted with contouring and polishing discs (Super-Snap Rainbow Technique Kit, SHOFU). Then proximal surfaces were polished using proximal sandpaper strips. Occlusion was checked for premature contacts. Two calibrated observers who were blinded to the objective of this study performed the evaluations. Color match, marginal adaptation, marginal discoloration, anatomic form, retention, secondary caries, and gloss retention were the properties evaluated for the restorations at baseline, 6, 12, 24, and 36 months using Modified Ryge Criteria (USPHS Criteria). Data were evaluated using the Chi-Square and Fisher's Exact tests (p=0.05).

ELIGIBILITY:
Inclusion Criteria:

* Being healthy without any chronic disease
* Having diastema, peg lateral or enamel defect in the anterior teeth
* Not having an occlusal anomaly such as bruxism or anterior crossbite
* Having a good oral hygiene
* Agreeing to come to the recall sessions regularly for 18 months
* Being over the age of 18

Exclusion Criteria:

* Having uncontrolled parafunction such as bruxism or anterior deep bite
* Having insufficient oral hygiene
* Being pregnant
* Having a systemic disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Marginal discoloration of prefabricated and resin composite veneers | 3 years
  Evaluating differently veneer options on anterior teeth with United State Public Health Service criteria regarding marginal discoloration by 2 independent evaluators Marginal discolouration was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth.
  Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth.
  Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction.
Marginal adaptation of prefabricated and resin composite veneers | 3 years
  Evaluating differently veneer options on anterior teeth with United State Public Health Service criteria regarding marginal adaptation by 2 independent evaluators Marginal discolouration was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth.
  Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth.
  Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction.
Retention rates of prefabricated and resin composite veneers | 3 years
  Evaluating differently veneer options on anterior teeth with United State Public Health Service criteria regarding retention rates by 2 independent evaluators Marginal discolouration was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth.
  Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth.
  Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction.
Anatomic form of prefabricated and resin composite veneers | 3 years
  Evaluating differently veneer options on anterior teeth with United State Public Health Service criteria regarding anatomic form by 2 independent evaluators Marginal discolouration was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth.
  Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth.
  Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction.
Color changes of prefabricated and resin composite veneers | 3 years
  Health Service criteria regarding color changes by 2 independent evaluators Marginal discolouration was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth.
  Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth.
  Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University School of Dentistry Department of Restorative, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No